CLINICAL TRIAL: NCT02946554
Title: Multicenter Phase II Safety and Preliminary Efficacy Study of 2 Dose Regimens of HepaStem in Patients With Acute on Chronic Liver Failure
Brief Title: Phase II Safety Study of 2 Dose Regimens of HepaStem in Patients With ACLF
Acronym: HEP101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellaion SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEP101
Record Dates: First submitted 2016-10-13; First posted 2016-10-27 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: Acute-On-Chronic Liver Failure; ACLF
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose cohort (Other): Two dose regimens of HepaStem will be given, which differ in the amount of cells per infusion.
  The low dose regimen will be given to the first cohort (first 6 patients included in the study).
  Interventions: Biological: HepaStem
- High dose cohort (Other): The high dose regimen will be given to the second cohort after evaluation of the safety of the 1st cohort (stepwise approach)
  Interventions: Biological: HepaStem

INTERVENTIONS:
Biological: HepaStem

SUMMARY:
The study will assess the safety of different dose regimens of HepaStem in cirrhotic Patients with ACLF or with acute decompensation at risk of developing ACLF up to Day 28 of the active study period.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosed cirrhosis
* Patient with Acute Decompensation of cirrhosis
* Serum total Bilirubin ≥ 6 mg/dL (≥100 umol/L)
* The INR measurement has to be : 1.2 ≤ INR < 2

Main Exclusion Criteria:

* Absence of portal vein flow
* Known or medical history of thrombotic events
* Gastrointestinal hemorrhage requiring blood transfusion
* Variceal bading or sclerosis within 4 weeks before infusion
* Septic shock or non-controlled bacterial infection
* Clinical evidence of aspergilus infection.
* Circulatory failure
* Respiratory disordered
* Coagulation disorders defined as INR ≥ 2, Fibrinogen < 100 mg/dL or Platelets < 50.000/mm3
* MELD score > 30.
* Major invasive procedure within 4 weeks before infusion
* Previous organ transplantation and/or ongoing immunosuppressive treatments.
* Renal failure due to chronic kidney disease.
* Clinically significant left-right cardiac shunt.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Safety assessed by occurence of Adverse Events (AE) up to Day 28 of the active study period | up to 28Day post first infusion day

SECONDARY OUTCOMES:
Efficacy assessed by clinical parameters | 28Day, 3 month and 1 year post first infusion day
  Clinical efficacy parameters evaluated by mortality, liver transplantation and disease scoring.
Efficacy assessed by biological parameters | 28Day, 3 month and 1 year post first infusion day
  Biological efficacy parameters evaluated by bilirubin, creatinine, INR and albumin values
Long term safety Follow up assessed by the occurence of Adverse Event of Special Interest | 3 month and 1 year post first infusion day
  Adverse Event of Special Interest defined as : SAE (Serious Adverse Event) with fatal

CONTACTS AND LOCATIONS:
Locations (10):
- Belgium (7):
  - CHU Brugmann, Brussels
  - Hôpital Erasme, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - KU Leuven, Leuven
  - CHU de Liège, Liège
  - Cliniques St Luc, Woluwe-Saint-Lambert
- France (3):
  - Hôpital Beaujon, Clichy
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Paul Brousse, Villejuif